CLINICAL TRIAL: NCT05566223
Title: A Phase 1/2 Trial (CheckCell-2) in Patients With Metastatic Non-small Cell Lung Cancer (NSCLC) Administering Tumor-Infiltrating Lymphocytes (TILs) in Which the Gene Encoding CISH Was Inactivated Using the CRISPR/Cas9 System
Brief Title: CISH Inactivated TILs in the Treatment of NSCLC
Acronym: CheckCell-2
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Intima Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2022LC001
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Metastatic Non Small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer; Squamous Cell Lung Cancer; Adenocarcinoma of Lung; Large Cell Lung Cancer
Keywords: PD-L1 negative; PD-L1 positive; Adoptive Cell Therapy; Immunotherapy; Gene Therapy; CISH Checkpoint; CRISPR; Gene Edit
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; aldesleukin; Interleukin-2; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CISH CRISPR TIL / Phase I Arm (Experimental): Dose Escalation/Expansion Cohort
  Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine +escalating doses of CISH inactivated TIL + high-dose aldesleukin
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: CISH Inactivated TIL; Drug: Aldesleukin
- CISH CRISPR TIL plus pembrolizumab / Phase I Arm (Experimental): Dose Expansion with Maintenance Therapy Cohort
  Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine +escalating doses of CISH inactivated TIL + high-dose aldesleukin
  Maintenance pembrolizumab during follow-up
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: CISH Inactivated TIL; Drug: Aldesleukin; Drug: Pembrolizumab
- CISH CRISPR TIL / Phase II Arm PD-L1 Negative Cohort (Experimental): Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine +recommended phase II dose (from phase I) of CISH inactivated TIL + high-dose aldesleukin
  May include maintenance pembrolizumab during follow-up
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: CISH Inactivated TIL; Drug: Aldesleukin; Drug: Pembrolizumab
- CISH CRISPR TIL / Phase II Arm PD-L1 Positive Cohort (Experimental): PD-L1 positive is defined as tumors with a PD-L1 Tumor Proportion Score (TPS) ≥ 1%.
  Non-myeloablative, lymphodepleting preparative regimen of cyclophosphamide and fludarabine +recommended phase II dose (from phase I) of CISH inactivated TIL + high-dose aldesleukin
  May include maintenance pembrolizumab during follow-up
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Biological: CISH Inactivated TIL; Drug: Aldesleukin; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Fludarabine — Day -7 to Day -3 : Fludarabine 25 mg/m^2/dose as a 1 hour intravenous infusion per institutional guidelines once a day for 5 doses beginning on Day -7. Fludarabine will be started approximately 1 to 2 hours after the cyclophosphamide on Day -6 and Day -5.
  Other Names: Fludara
Drug: Cyclophosphamide — Day -6 and Day -5: Cyclophosphamide 60 mg/kg/dose as a 2 hour intravenous infusion with Mesna 15 mg/kg/dose, 1st dose prior to Cyclophosphamide infusion then at 3,6,9 and 12 hours later.
  Other Names: Cytoxan
Biological: CISH Inactivated TIL — Day 0 : Each bag of autologous CISH inactivated TIL for infusion will be administered intravenously (IV) on the Patient Care Unit over 10-20 minutes at assigned dose level.
Drug: Aldesleukin — Days 1-4 : Aldesleukin at 720,000 U/kg as an intravenous infusion, every 8 -12 hours but, no more than 24 hours apart as tolerated for up to 6 doses.
  Other Names: Proleukin; Interleukin-2; IL-2
Drug: Pembrolizumab — Administered as maintenance therapy in some patients starting at first follow-up (400 mg/dose starting Day 28 /Week 4 then every 6 weeks thereafter until disease progression, unacceptable toxicity, or up to 24 months)
  Other Names: Keytruda
  Arms: CISH CRISPR TIL / Phase II Arm PD-L1 Negative Cohort; CISH CRISPR TIL / Phase II Arm PD-L1 Positive Cohort; CISH CRISPR TIL plus pembrolizumab / Phase I Arm

SUMMARY:
A clinical trial to assess the safety and efficacy of genetically-engineered Tumor Infiltrating Lymphocytes (TIL) in which the intracellular immune checkpoint CISH has been inhibited using CRISPR gene editing for the treatment of Metastatic Non-small Cell Lung Cancer (NSCLC).

DETAILED DESCRIPTION:
Tumor Infiltrating Lymphocytes (TIL) have shown efficacy in certain cancers, principally in melanoma, but also in non-small cell lung cancer (NSCLC). Combination cell surface checkpoint inhibitor therapy has also been employed in an attempt to enhance the efficacy of these cell therapies. Genetic engineering of T cells to further increase anti-tumor activity is now possible.

CISH (Cytokine-induced SH2 protein) is a novel intra-cellular immune checkpoint and an important negative regulator of T-cell signaling and function. The inhibition of CISH in mouse anti-tumor lymphocytes results in a marked increase in the ability of these lymphocytes to mediate tumor regression following administration to tumor bearing mice.

Additionally, data in genetically-engineered, neoantigen-specific human T cells in which CISH was inhibited, showed enhanced TCR functional avidity and increased ability of these T cells to detect cancer specific mutations and mount robust polyfunctional cytokine immune responses against their cognate cancer antigens. Thus, these T cells appear to have a significant advantage in inducing anti-tumor responses compared to wild-type anti-tumor lymphocytes.

The researchers have developed and optimized a CRISPR/Cas9 based strategy for precise and efficient genetic engineering in primary human T-cells without sacrificing cell viability or function, allowing for inhibition of a heretofore undruggable intracellular checkpoint.

Thus, in this protocol, the researchers propose to inhibit the gene encoding the intracellular checkpoint target CISH in TIL from patients with metastatic NSCLC whose tumors are PD-L1 negative or positive in order to evaluate the safety and efficacy of genetically engineered T cell therapy in the setting of novel checkpoint inhibition .

ELIGIBILITY:
Inclusion Criteria (1st Screening prior to Tumor Resection - See below for evaluation of continuing eligibility prior to start of investigational treatment):

* Confirmed histologic diagnosis of either PD-L1 negative or positive metastatic non-small cell lung cancer (NSCLC)
* Candidate to receive 1st line treatment with anti-PD-1/anti-PD-L1 immunotherapy in combination with chemotherapy or be within 6 months (Phase 1) or 3 months (Phase 2) of initiation of this type of systemic treatment (regardless of where such treatment was started) when the tumor resection is performed. Patients who have received adjuvant or neoadjuvant anti-PD-1/anti-PD-L1 immunotherapy and/or chemotherapy can be screened for the trial if they experienced a relapse more than 6 months from the end of their last systemic treatment. The tumor resection for investigational product manufacturing should be undertaken before the initiation of this 1st line therapy; however, patients who have already started their 1st line treatment should have these procedures performed and completed as soon as deemed clinically appropriate, but no later than 6 months (Phase 1) or 3 months (Phase 2) from the start of 1st line treatment. After documented radiographic disease progression on or following this 1st line of treatment, patients will receive investigational product as 2nd line therapy.
* Measurable disease per RECIST v1.1 with at least one lesion identified as resectable for cell therapy manufacturing (minimum volume of tumor tissue required is 1 cm^2 as single mass or fragments) and at least one other lesion meeting the RECIST criteria for measurable disease to serve as an indicator of disease response. The location of the tumor resection and method used to obtain tumor (i.e., laparoscopy, endoscopic ultrasound, etc.) will be determined based on an individual patient's disease. Note: previously irradiated lesions with radiographic progression are not eligible for tumor resection.
* Patients who have asymptomatic and or treated brain metastases are eligible, but must be discussed with and approved by the Coordinating Investigator. Lesions that have been treated with stereotactic radiosurgery must be clinically stable for 1 month after treatment for the patient to be eligible. Patients with surgically resected brain metastases are eligible. Patients with brain metastases must not be receiving systemic steroids (oral progestin/estrogen combinations used for contraception are an exception). Brain metastases are assessed using the RANO-BM criteria.
* Clinical performance status of Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1 and an estimated life expectancy of ≥ 6 months.
* Age ≥ 18 years and ≤ 70 years.
* Hematology within 14 days of study enrollment:

  * Absolute neutrophil count > 1000/mm^3 without the support of filgrastim
  * White Blood Cells (WBC) ≥ 3000/mm^3
  * Platelet count ≥ 75,000/mm^3
  * Hemoglobin > 8.0 g/dL. Subjects may be transfused to reach this cutoff.
* Adequate organ function within 14 days of study enrollment defined as:

  * Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 5.0 x upper limit of normal (ULN)
  * Serum creatinine ≤ 1.6 mg/dL or creatinine clearance by Cockroft-Gault ≥ 50 mL/min.
  * Total bilirubin ≤ to 2.0 mg/dL, except in patients with Gilbert's Syndrome, who must have a total bilirubin ≤ 3.0 mg/dL.
* Serology testing within 3 months of study enrollment (tumor resection):

  * Seronegative for HIV antibody. (The investigational treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immunocompetence and thus may be less responsive to the study treatment and more susceptible to its toxicities.)
  * Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.
* Sexually active females of childbearing potential and males with female partners of childbearing potential must agree to use effective contraception for the duration of study treatment starting with Screening and for 12 months (females) and 4 months (males) after the last dose of cyclophosphamide; if receiving pembrolizumab, for 4 months (females and males) after the last dose of pembrolizumab. Examples of effective contraception include oral progestin/estrogen combinations (an exception to the strict prohibition of systemic steroid use), an IUD or implant plus a condom. Women of non-childbearing potential are defined as those who have no uterus, ligation of the fallopian tubes, or permanent cessation of ovarian function due to ovarian failure or surgical removal of the ovaries. A woman also is presumed to be infertile due to natural causes if she has been amenorrheic for > 12 months and/or has a follicle-stimulating hormone (FSH) > 40 IU/L.
* Agrees to remain near the treatment site (within approximately a 1-hour drive) after the investigational product infusion through the Day 28/Week 4 follow-up visit.
* Voluntary written consent prior to the performance of any research-related procedures.

Exclusion Criteria (1st Screening prior to Tumor Resection - See below for evaluation of continuing eligibility prior to start of investigational treatment):

* Known oncogene driver mutations (e.g., including but not limited to, epidermal growth factor receptor [EGFR], anaplastic lymphoma kinase [ALK], reactive oxygen species [ROS], Kirsten RAt Sarcoma Virus G12C [KRAS G12C], human epidermal growth factor receptor 2 [HER2], neurotrophic tyrosine receptor kinase [NTRK], BRAF V600E, RET fusion positive, mesenchymal-epithelial transition gene exon 14 [METex14]) which are sensitive to targeted Food and Drug Administration (FDA)-approved therapies.
* Pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant. Women of childbearing potential must have a negative pregnancy test (serum or urine) within 7 days of enrollment.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* Prior treatment with any cell therapy product or organ allograft within the past 20 years.
* Patients who have had another primary malignancy within the previous 3 years.
* Concurrent opportunistic infection.
* Receipt of a live or attenuated vaccination within 28 days prior to the tumor harvest.
* Active systemic infections requiring anti-infective treatment, coagulation disorders, or any other active major medical illnesses.
* Use of systemic steroids (0 mg) within 14 days prior to tumor collection or anticipated need of systemic steroids (0 mg) within 21 days prior to investigational product infusion or anticipated any time after that infusion (oral progestin/estrogen combinations used for contraception are an exception).
* History of severe immediate hypersensitivity reaction to cyclophosphamide, fludarabine, aldesleukin, pembrolizumab, or dimethyl sulfoxide (DMSO).
* History of coronary revascularization or ischemic symptoms, myocarditis, congestive heart failure (as defined by New York Heart Association Functional Classification III or IV), serious uncontrolled cardiac arrhythmia, or other clinically significant cardiac disease that may increase the risk associated with study participation, in the opinion of the investigator.
* Documented left ventricular ejection fraction (LVEF) ≤ 45%.
* History of Grade ≥ 2 pneumonitis or active interstitial lung disease/pneumonitis requiring treatment with systemic steroids.
* Documented forced expiratory volume in 1 second (FEV1) ≤ 50% or FEV1/forced vital capacity (FVC) ≤ 0.7 (6-minute walk test if unable to perform or unreliable spirometry).
* Clinically significant patient history that, in the judgment of the enrolling investigator, would compromise the patient's ability to tolerate high-dose aldesleukin.
* Receiving any investigational agents within 21 days prior to tumor collection.
* Medical status or social situation that may make study participation not in the best interest of the patient in the opinion of the enrolling investigator.

Criteria for Confirmation of Continuing Eligibility (2nd Screening Prior to Hospital Admission for Investigational Treatment Start)

* Measurable disease per RECIST v1.1 within 4 weeks of starting lymphodepleting chemotherapy.
* Clinical performance status of ECOG 0 or 1.
* Adequate hematologic, liver, and renal laboratory parameters within 7 days of starting lymphodepleting chemotherapy:

  * Absolute neutrophil count > 1000/mm^3 without the support of filgrastim
  * WBC ≥ 3000/mm^3
  * Platelet count ≥ 75,000/mm^3
  * Hemoglobin > 8.0 g/dL. Subjects may be transfused to reach this cutoff.
  * Serum ALT and AST ≤ 5.0 x ULN
  * Serum creatinine ≤ 1.6 mg/dL or creatinine clearance by Cockroft-Gault ≥ 50 mL/min.
  * Total bilirubin ≤ to 2.0 mg/dL, except in patients with Gilbert's Syndrome, who must have a total bilirubin ≤ 3.0 mg/dL.
* Seronegative for HIV antibody, HbsAg, anti-HBc, and hepatitis C antibody as tested within 3 months of beginning lymphodepleting chemotherapy. If anti-HBc is positive, patient must have negative HBV DNA to be eligible. Seronegative for anti-HCV. If anti-HCV test is positive, then patient must be tested for HCV by RT-PCR and be HCV RNA negative.
* Negative SARS-CoV-2 by RT-PCR or antigen test within 7 days of starting lymphodepleting chemotherapy.
* More than 4 weeks must have elapsed since the last dose of prior systemic therapy and the start of the lymphodepleting chemotherapy, and acute toxicities must have recovered to Grade 1 or less (except for toxicities such as alopecia or vitiligo). Minor surgical procedures within the 3 weeks prior to of the start of lymphodepleting chemotherapy is permitted as long as all toxicities have recovered to Grade 1 or less.
* Continues to agree to use of contraception for sexually active females of childbearing potential and males with female partners of childbearing potential.
* Negative pregnancy test within 7 days of starting lymphodepleting chemotherapy in women of childbearing potential.
* No concurrent opportunistic infection.
* No receipt of a live or attenuated vaccination within 28 days prior to the start of lymphodepleting chemotherapy.
* No active systemic infections requiring anti-infective treatment, coagulation disorders, or any other active major medical illnesses.
* No requirement for or use of systemic steroids (0 mg) within 21 days prior to investigational product infusion or anticipated any time after that infusion (oral progestin/estrogen combinations used for contraception are an exception).
* 13. No history of coronary revascularization or ischemic symptoms, myocarditis, congestive heart failure (as defined by New York Heart Association Functional Classification III or IV), serious uncontrolled cardiac arrhythmia, or other clinically significant cardiac disease that may increase the risk associated with study participation in the opinion of the investigator.
* If ≥ 12 weeks has passed since initial screening test or if clinically indicated, confirm LVEF is not ≤ 45%.
* No history of Grade ≥ 2 pneumonitis or active interstitial lung disease/pneumonitis requiring treatment with systemic steroids.
* If ≥ 12 weeks has passed since initial screening test or if clinically indicated, confirm FEV1 is not ≤ 50% or FEV1/FVC is not ≤ 0.7 (6 minute walk test if unable to perform or unreliable spirometry).
* No change in medical status or social situation that would make study participation not in the best interest of the patient in the opinion of the enrolling investigator.
* Continues to agree to remain near the site (within approximately a 1-hour drive) after the investigational product infusion through the Day 28 /Week 4 follow-up visit.
* Agrees to and signs the consent form for the LTFU study (2022LC LTFUP 001).
* Voluntarily signed the study treatment consent form within 28 days prior to the start of the lymphodepleting chemotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Phase I: Safety and Initial Efficacy | 11 months
  Safety by type, incidence, severity, seriousness, and relation of study treatment of AEs, DLTs, and laboratory abnormalities. Initial efficacy per RECIST v1.1
Phase II: Objective Response Rate (ORR) | 3.5 years
  RECIST v1.1

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 2-5 years
  Kaplan-Meier estimate
Overall Survival (OS) | 2-5 years
  Kaplan-Meier estimate
Duration of Response (DoR) | 2-5 years
  Length of time that target lesion(s) continue to respond to treatment without growing or spreading
Clinical Benefit Rate | 2-5 years
  Percentage of combined patients who achieve complete response, partial response and stable disease
Tumor Growth Change | 2-5 years
  Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used in the RECIST v1.1 criteria
Toxicity Incidence | 2-5 years
  Incidence of targeted toxicities events

CONTACTS AND LOCATIONS:
Overall Officials: Emil Lou, MD, PhD, Principal Investigator — Division of Hematology, Oncology, and Transplantation, University of Minnesota; Erminia Massarelli, MD, PhD, MS, Principal Investigator — Department of Medical Oncology & Therapeutics Research, City of Hope
Locations (2):
- United States (2):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota